CLINICAL TRIAL: NCT03757377
Title: Clinical Evaluation of Safety and Effectiveness of the BackBeat Medical Moderato System in Patients With Hypertension: A Double-Blind Randomized Trial
Brief Title: Moderato System in Patients With Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BackBeat Medical Inc (Industry)
Collaborators: Massachusetts General Hospital (Other); MLM Medical Labs GmbH (Industry); nabios GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS-03 Ver 3.0
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Hypertension, Resistant to Conventional Therapy; Atrioventricular Block
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BackBeat Moderato System (PHC ON) (Active Comparator): Eligible patients randomized after optimization phase to PHC ON (PHC algorithm active) for 12 months. Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator.
  Interventions: Device: BackBeat Moderato System
- BackBeat Moderato System (PHC OFF) (Placebo Comparator): Eligible patients randomized after optimization phase to pacemaker only (PHC OFF or PHC algorithm not active) for 12 months. Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator.
  Interventions: Device: BackBeat Moderato Sytsem

INTERVENTIONS:
Device: BackBeat Moderato System — Eligible patients randomized after optimization phase to PHC ON for 12 months. Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator
  Arms: BackBeat Moderato System (PHC ON)
Device: BackBeat Moderato Sytsem — Eligible patients randomized after optimization phase to PHC OFF for 12 months. Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator.
  Arms: BackBeat Moderato System (PHC OFF)

SUMMARY:
The purpose of this double blind randomized study is the evaluation of the safety and efficacy of the Moderato System. The Moderato implantable pulse generator is indicated for patients who have hypertension and also require a dual chamber pacemaker in order to reduce their blood pressure.

In this amended CS-03 protocol Version 3.0, the study will evaluate the safety and efficacy in a randomized, double-blind study following active treatment vs. a control patient population for a period of 3 month for efficacy and 12 months for safety (In comparison to 6 months for patients under protocol CS-03 Ver 1.1, NCT02837445).

The device will be considered to have a clinical effectiveness with regard to its anti-hypertension function if there is a statistically significant and clinically meaningful reduction in mean 24-hour ambulatory systolic blood pressure in the treatment group compared to the control group. The primary efficacy endpoint will be evaluated 3 months after randomization. The Primary safety analysis will compare the treatment and the control after 12 months of treatment.

DETAILED DESCRIPTION:
Protocol CS-03 Ver 1.1 (NCT02837445) was amended at the advice of the Scientific Advisory to protocol CS-03 Version 3.0 with more stringent hypertension inclusion criteria and different observation intervals for efficacy and safety.

In CS-03 Version 3.0 the time of the primary efficacy endpoint was reduced from 6 months to 3 months post randomization which was deemed a suitable interval for the chronic effect, whereas for the safety endpoint, the period was lengthened to 12 months post randomization to better monitor potential risks of the treatment on cardiac function (Blinding period was increased from 6 months to 12 months). Protocols were thus split in order to allow better clarification to the difference in the time to the primary endpoints for efficacy and safety between the two CIP versions and simplify data analysis.

Protocol Ver 3.0 prescribes data analysis of all patients randomized under version 1.1 to be performed once they complete the 6 months follow-up as set in protocol version 1.1 (NCT0283744). It is expected that ~40 patients will be randomized according to protocol version 1.1 prior to the enrollment of patients according to protocol version 3.0. The results will be considered as interim analysis.

The recruitment for the protocol version 1.1 is now completed. Total of 47 patients were randomized according to protocol version 1.1 and all patients completed the follow-up period for the primary endpoint.

Patients are currently being followed up for the study "extension period".

ELIGIBILITY:
Inclusion Criteria:

* Requirement of dual chamber pacemaker or upgrade from a single chamber to a dual chamber pacemaker.
* Stable (at least 6 weeks) hypertension treatment with at least 1 anti-hypertensive drug, which is anticipated to be maintained without changes. Stable is defined as being in the same drug regimen, and the dose of each drug(s) no more than 50% reduced or 100% increased over the past 6 weeks.
* Average 24-hour ambulatory systolic blood pressure ≥ 130 mmHg (with directly observed medical therapy, DOT) and office blood pressure ≥140 mmHg.
* Subject is able to comply with study visits for at least 13 months (e.g., is capable and willing to travel to/from the center for all scheduled study visits).

Exclusion Criteria:

* Known secondary cause of HTN.
* Average ambulatory or office systolic BP > 195 mmHg.
* Permanent atrial fibrillation.
* History of significant paroxysmal atrial fibrillation/flutter burden (defined as >25% of beats).
* Cardiac ejection fraction <50%.
* Symptoms of heart failure, NYHA Class II or greater.
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy or inter-ventricular septal thickness ≥ 15 mm.
* Subject is on dialysis.
* Subject has an estimated Glomerular Filtration Rate < 30 ml/min/1.73 m²
* Prior neurological events (stroke or TIA) within the past year or events at a prior time that has resulted in residual neurologic deficit.
* Carotid artery disease.
* Known autonomic dysfunction.
* History of clinically significant untreated ventricular tachyarrhythmia or has experienced cardiac arrest.
* Previous active device-based treatment for HTN.
* Existing implant, other than a pacemaker that needs replacing.
* Subject is or has the possibility of becoming pregnant and is unwilling of contraception during the study.
* Subject is unwilling or cannot provide Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of composite of major cardiac events | 12 months post Randomization
  including heart failure, clinically significant arrhythmias eg, persistent or increased atrial fibrillation, serious ventricular arrhythmias, myocardial infarction, stroke, heart failure, renal failure and/or related safety events that result in death
Change in average 24 hour systolic ambulatory blood pressure | Week 3 pre Randomization and 3 months post Randomization

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof. MD, Principal Investigator — Asklepios Klinik St. Georg
Locations (4):
- UZ Brussel - Heart Rhythm Management Center, Brussels, Belgium
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania
- Poland (2):
  - Samodzielnym Publicznym Centralnym Szpitalem Klinicznym, Warsaw
  - Silesian Center for Heart Diseases, Zabrze

REFERENCES:
- See also: Rationale and evidence for the development of a durable device-based cardiac neuromodulation therapy for hypertension. — https://www.ncbi.nlm.nih.gov/pubmed/?term=29628351
- See also: Pacemaker-Mediated Programmable Hypertension Control Therapy. — https://www.ncbi.nlm.nih.gov/pubmed/?term=29275370